CLINICAL TRIAL: NCT01960751
Title: Etude Des Séquelles Neurocognitives À Long Terme Des Faibles Doses De Radiation Chez 150 Patients Traités Par Radiothérapie Dans L'enfance Pour Un Hémangiome Cutané À L'Institut Gustave Roussy (IGR) Entre 1941 Et 1973
Brief Title: Long Term Neurocognitive Effects of Low-dose Radiation in the Brain: Study of 150 Patients in the French Hemangioma Cohort
Acronym: CogRad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: European Commission (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: C13-01; 2013-A00513-42 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-08-07; First posted 2013-10-11 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Patients Treated by Radiotherapy with < One Gy to the Brain
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neurocognitive tests (Other): neurocognitive tests battery (MMSE, SDS, SF-36, HAD, BPRS, RAVLT, FACT-Cog, MoCA)
  Interventions: Other: neurocognitive tests battery

INTERVENTIONS:
Other: neurocognitive tests battery — The two groups (exposed: 0.05 to 1 Gy; unexposed: less than 0.05 Gy) will receive the same neurocognitive tests battery.
  Other Names: - MMSE; - SDS; - SF-36; - HAD; - BPRS; - RAVLT; - FACT-Cog; - MoCA

SUMMARY:
Context: Studies that address specifically the neurocognitive consequences that can be caused by low-dose radiation receiving during the childhood have still to be performed. In this issue, we focus on an investigation with patients who have received radiotherapy for a benign tumor (skin hemangioma), in France.

Patients and methods: More than 8300 children with a skin hemangioma were treated at Gustave Roussy (Île-de-France) from 1941 to 1973 and a number of them have received radiotherapy. These patients have been treated and followed by Gustave Roussy, so their clinical records can be tracked with great accuracy and the ionizing radiation dose to the brain have been estimated. From this patient cohort, the aim is to evaluate neurocognitive dysfunction or disorder that can be caused by low-dose radiation to the brain (less than one Gray (Gy)). A total of 150 patients is expected. They will be contacted by letter to explain the purpose and methods of carrying out tests. Two groups will be analysed according to the received ionizing radiation dose to the brain during the radiotherapy (exposed: 0.05 to 1 Gy, vs unexposed: less than 0.05 Gy). Tests exploring several cognitive functions (memory, arithmetic, orientation, etc.) will be used.

Expected results: We expect to describe the potential neurocognitive dysfunction or disorder and to identify risk factors and brain structures whose lesions are responsible for the neurocognitive dysfunction or disorder.

A therapeutic treatment will be proposed in the eventuality of screening of a neurocognitive dysfunction or disorder.

DETAILED DESCRIPTION:
CogRad is an interventional study designed within the European project called Cognitive and Cerebrovascular Effects Induced by Low Dose Ionizing Radiation (CerebRad).

CerebRad is a collaborative European project funded in 2011 within the 7th European Union (EU) framework programme, Nuclear Fission and Radiation Protection. CerebRad aims to identify the potential cognitive and cerebrovascular risks of radiation doses below 100 milliGray (mGy) when delivered to a young child (pre- or postnatally).

ELIGIBILITY:
Inclusion Criteria:

* Subject treated by radiotherapy for a skin hemangioma in childhood at Gustave Roussy between 1941 and 1973 and who have received less than 1 Gy of radiation doses in the brain
* Inhabitants of Île-de-France
* French medical insurance
* Good knowledge and understanding of the French language

Non-inclusion Criteria

* Cerebral hemangioma
* Syndrome genetic predisposition
* Pregnant woman
* Private person of liberty or under guardianship
* Radiation dose to the brain greater than 1 Gy during radiotherapy treatment of skin hemangioma
* Chemotherapy during skin hemangioma treatment
* Inability to undergo counseling for geographical reasons

Exclusion Criteria:

* Pregnancy
* Inability to perform neurocognitive tests battery for medical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-04-14 (Actual); Primary Completion 2015-02-04 (Actual); Study Completion 2015-02-04 (Actual)

PRIMARY OUTCOMES:
All neurocognitive dysfunction or disorder on adults measured by means of eight tests | Participants will be tested for the duration of hospital stay (half a day).The neurocognitive tests battery will be carry out 56 years on average after exposure to low-dose radiation.
  The score to the 8 tests will be correlate with the presence of neurocognitive dysfunction or disorder

CONTACTS AND LOCATIONS:
Overall Officials: Chiraz EL-FAYECH, Study Director — Gustave Roussy, France; Florent DE VATHAIRE, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Gustave Roussy, Villejuif, France

REFERENCES:
- [Background] Fragu P, Lemarchand-Venencie F, Benhamou S, Francois P, Jeannel D, Benhamou E, Sezary-Lartigau I, Avril MF. Long-term effects in skin and thyroid after radiotherapy for skin angiomas: a French retrospective cohort study. Eur J Cancer. 1991;27(10):1215-22. doi: 10.1016/0277-5379(91)90084-q. PMID 1835589
- [Background] Ron E, Modan B, Boice JD Jr, Alfandary E, Stovall M, Chetrit A, Katz L. Tumors of the brain and nervous system after radiotherapy in childhood. N Engl J Med. 1988 Oct 20;319(16):1033-9. doi: 10.1056/NEJM198810203191601. PMID 3173432
- [Background] Little MP, Hawkins MM, Shore RE, Charles MW, Hildreth NG. Time variations in the risk of cancer following irradiation in childhood. Radiat Res. 1991 Jun;126(3):304-16. PMID 2034788
- [Background] Hall P, Adami HO, Trichopoulos D, Pedersen NL, Lagiou P, Ekbom A, Ingvar M, Lundell M, Granath F. Effect of low doses of ionising radiation in infancy on cognitive function in adulthood: Swedish population based cohort study. BMJ. 2004 Jan 3;328(7430):19. doi: 10.1136/bmj.328.7430.19. PMID 14703539
- [Background] Haddy N, Andriamboavonjy T, Paoletti C, Dondon MG, Mousannif A, Shamsaldin A, Doyon F, Labbe M, Robert C, Avril MF, Fragu P, Eschwege F, Chavaudra J, Schvartz C, Lefkopoulos D, Schlumberger M, Diallo I, de Vathaire F. Thyroid adenomas and carcinomas following radiotherapy for a hemangioma during infancy. Radiother Oncol. 2009 Nov;93(2):377-82. doi: 10.1016/j.radonc.2009.05.011. Epub 2009 Jun 8. PMID 19515442
- [Background] Haddy N, Mousannif A, Paoletti C, Dondon MG, Shamsaldin A, Doyon F, Avril MF, Fragu P, Labbe M, Lefkopoulos D, Chavaudra J, Robert C, Diallo I, de Vathaire F. Radiotherapy as a risk factor for malignant melanoma after childhood skin hemangioma. Melanoma Res. 2012 Feb;22(1):77-85. doi: 10.1097/CMR.0b013e32834dcff1. PMID 22082956
- [Background] Haddy N, Dondon MG, Paoletti C, Rubino C, Mousannif A, Shamsaldin A, Doyon F, Labbe M, Robert C, Avril MF, Demars R, Molinie F, Lefkopoulos D, Diallo I, de Vathaire F. Breast cancer following radiotherapy for a hemangioma during childhood. Cancer Causes Control. 2010 Nov;21(11):1807-16. doi: 10.1007/s10552-010-9607-5. Epub 2010 Jul 7. PMID 20607383
- [Background] Dondon MG, de Vathaire F, Shamsaldin A, Doyon F, Diallo I, Ligot L, Paoletti C, Labbe M, Abbas M, Chavaudra J, Avril MF, Fragu P, Eschwege F. Cancer mortality after radiotherapy for a skin hemangioma during childhood. Radiother Oncol. 2004 Jul;72(1):87-93. doi: 10.1016/j.radonc.2004.03.011. PMID 15236880
- [Background] Ligot L, Diallo I, Shamsaldin A, Chavaudra J, BonaIti-Pellie C, de Vathaire F. Individualized phantom based on CT slices and auxological data (ICTA) for dose estimations following radiotherapy for skin haemangioma in childhood. Radiother Oncol. 1998 Dec;49(3):279-85. doi: 10.1016/s0167-8140(98)00099-1. PMID 10075261